CLINICAL TRIAL: NCT02942498
Title: Clinical Trials Phase III, Double Blind, Crossover to Asses the Safety and Efficacy of Vitamin C and Vitamin E in Combination Versus Placebo for Treating Cognitive and Behavior Disorder in Children With Fragile X Syndrome
Brief Title: Clinical Trial for Asses the Safety and Efficacy of Vitamin C and Vitamin E in Combination Versus Placebo for Treating Cognitive and Behavior Disorder in Children With Fragile X Syndrome
Acronym: SXF2-8
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Collaborators: Delos Clinical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SXF2-8
Record Dates: First submitted 2016-10-07; First posted 2016-10-24 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2016-09

CONDITIONS: X Fragile Syndrome
Keywords: behavior, cognitive
MeSH Terms: conditions — Fragile X Syndrome; Behavior | interventions — Ascorbic Acid; Vitamin E

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin C 10 mg/Kg + Vitamin E 10 mg/Kg (Experimental): Vitamin C and Vitamin E supplementation 10 mg/kg/ day
  Interventions: Drug: Vitamin C 10mg/Kg Vitamin E 10 mg/Kg
- Placebo (Placebo Comparator): Placebo solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin C 10mg/Kg Vitamin E 10 mg/Kg
  Arms: Vitamin C 10 mg/Kg + Vitamin E 10 mg/Kg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine vitamin C and vitamin E in combination are effective in the treatment of cognitive and behavior disorder in children with fragile X syndrome.

DETAILED DESCRIPTION:
The combination of vitamin E and vitamin C supplementation has been associated with a lower prevalence (-78%) and incidence (-64%) of Alzheimer's disease in the elderly population. It has recently been shown that dietary vitamin E supplementation reduces the production of free radicals inhibiting NADPH oxidase activity in circulating neutrophils. Another work describes the inhibition of glutamate release by activated microglia in cell cultures incubated with vitamin E, effect that can prevent excitotoxicity.

The investigators propose to evaluate the effectiveness of treatment in neurodevelopmental disorders affected by fragile X syndrome (FXS) with lipophilic compounds antioxidants such as tocopherol and hydrophilic compounds antioxidants such as ascorbic acid, which regulate oxidative stress and improve learning and behavioral mouse model and humans.

Our group has positive results in the use of this combination of antioxidants as a treatment for fragile X syndrome in adolescents. This disease has developed previous clinical trials with EUDRACT codes: 2009-017837-23 and 2013-004276-35.

The use of the combination of vitamin C and E in the treatment of cognitive and behavioral disorder in FXS, is patented PCT-050 187 with reference number 2011070875

This combination will be administered as a single oral dose with a total dose of 10mg / kg / day for each of the vitamins. This dose is maintained within the therapeutic range of both antioxidants.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Fragile X syndrome by genetic testing of molecular biology, full mutation result methylation.
2. Having an older age of 1 year and less than 9 years
3. Having signed the informed consent document before starting their participation in the trial.

Exclusion Criteria:

1. Any advanced, severe or unstable disease.
2. Individuals with other psychiatric diagnosis as the first diagnosis.
3. It have been suffered serious medical problems in the last 12 months.
4. Be taking more than 100 mg of vitamin E or C a day in the last month.
5. Having physical, mental or sensory impairments that prevent the assessment of effectiveness.
6. Hypersensitivity to any component of the preparation.
7. Liver failure or severe renal or previous history of kidney stones.
8. Any treatment regimen, including treatment with psychotropic drugs and / or anticonvulsant therapy that has not been stable for a period ≥ 4 weeks before randomization.
9. Current treatment with more than two psychoactive medications, excluding medication used specifically for the control of seizures.
10. Hypoprothrombinemia secondary to vitamin K deficiency
11. Sensitivity to any of the compounds of formula treatment.
12. Patients diagnosed with congenital or idiopathic methemoglobinemia for diagnosis of glucose-6-phosphate dehydrogenase deficiency.
13. Use of oral anticoagulants, iron or vitamin A.
14. Forecast initiate or change pharmacological or no pharmacological interventions during the course of the study.
15. Patients weighing less than 4.2 kg

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2016-07; Primary Completion 2017-09-25 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Autism Treatment Evaluation Checklist (ATEC). | 32 weeks
Global Clinical Impression (GCI) | 32 weeks
Peabody Picture Vocabulary Test (PiVT) | 32 weeks
Battelle developmental inventory screening | 32 weeks
Vineland Adaptive Behavior Scales | 32 weeks
Adverse event reported | 32 weeks
Quantitative Checklist for Autism in Toddlers (Q-Chat) test | 32 weeks

SECONDARY OUTCOMES:
Golberg scale GHQ-28 | 32 weeks
Quality life SF36 test | 32 weeks
Psychological General Well-Being Index | 32 weeks
Sleep Disturbance Scale for Children | 32 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Regional de Málaga, Málaga, Málaga, Spain

REFERENCES:
- [Background] Zandi PP, Anthony JC, Khachaturian AS, Stone SV, Gustafson D, Tschanz JT, Norton MC, Welsh-Bohmer KA, Breitner JC; Cache County Study Group. Reduced risk of Alzheimer disease in users of antioxidant vitamin supplements: the Cache County Study. Arch Neurol. 2004 Jan;61(1):82-8. doi: 10.1001/archneur.61.1.82. PMID 14732624
- [Background] Castilla P, Davalos A, Teruel JL, Cerrato F, Fernandez-Lucas M, Merino JL, Sanchez-Martin CC, Ortuno J, Lasuncion MA. Comparative effects of dietary supplementation with red grape juice and vitamin E on production of superoxide by circulating neutrophil NADPH oxidase in hemodialysis patients. Am J Clin Nutr. 2008 Apr;87(4):1053-61. doi: 10.1093/ajcn/87.4.1053. PMID 18400731
- [Background] Barger SW, Goodwin ME, Porter MM, Beggs ML. Glutamate release from activated microglia requires the oxidative burst and lipid peroxidation. J Neurochem. 2007 Jun;101(5):1205-13. doi: 10.1111/j.1471-4159.2007.04487.x. Epub 2007 Mar 30. PMID 17403030